CLINICAL TRIAL: NCT02980250
Title: A Clinical Multi-Center Study of Efficacy Analysis in Different Doses of Domperidone in Feeding Intolerance of Premature Infant
Brief Title: Multi-Center Study of Different Doses Domperidone in Feeding Intolerance
Acronym: MCSDDDFI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Guangdong Provincial Maternal and Child Health Hospital (Other); Shen-Zhen City Maternity and Child Healthcare Hospital (Other); Maternal and Child Health Hospital of Foshan (Other); Guangzhou Panyu Central Hospital (Other)
Responsible Party: Principal Investigator, Weimin Huang, The director of the neonatology department, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NFEC-2015-131
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Feeding Intolerance; Premature Birth; Domperidone Overdose; Gastric Retention
Keywords: feeding intolerance; premature infant; domperidone
MeSH Terms: conditions — Premature Birth | interventions — Contraceptives, Oral; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- low dose (Experimental): The premature infant in this group will be feed with 0.2mg/kg/tds domperidone suspension(motilium;100ml)for 7 days and will be tested the residual percentage everyday.
  Interventions: Drug: Low dose
- normal dose (Experimental): The premature infant in this group will be feed with 0.4mg/kg/tds domperidone suspension(motilium;100ml)for 7 days and will be tested the residual percentage everyday.
  Interventions: Drug: normal dose
- over dose (Experimental): The premature infant in this group will be feed with 0.6mg/kg/tds domperidone suspension(motilium;100ml)for 7 days and will be tested the residual percentage everyday.
  Interventions: Drug: over dose
- placebo (Placebo Comparator): The premature infant in this group will be feed with some vitamin which will dilute into the 5% glucose and have the same appearance and taste with the experimental team for 7 days and will be tested the residual percentage everyday.
  Interventions: Drug: Glucose

INTERVENTIONS:
Drug: Low dose — 0.2mg group-The premature infant will be fed with 0.2mg/kg/tds domperidone and will be tested the residual glucose everyday in a 7-days period.
  Other Names: Domperidone Suspension(Motilium), B12200018238
  Arms: low dose
Drug: normal dose — 0.4mg group-The premature infant will be fed with 0.4mg/kg/tds domperidone and will be tested the residual glucose everyday in a 7-days period.
  Other Names: Domperidone Suspension(Motilium), B12200018238
  Arms: normal dose
Drug: over dose — 0.6mg group-The premature infant will be fed with 0.6mg/kg/tds domperidone and will be tested the residual glucose everyday in a 7-days period.
  Other Names: Domperidone Suspension(Motilium), B12200018238
  Arms: over dose
Drug: Glucose — Glucose group-The premature infant will be fed with glucose and will be tested the residual glucose everyday in a 7-days period.
  Other Names: 5% Glucose
  Arms: placebo

SUMMARY:
The purpose of this clinical multi-center study is to determine whether different doses of domperidone are effective in the treatment of feeding intolerance in premature infant

DETAILED DESCRIPTION:
the premature infant have been divided into four group.The first group take the 0.2mg/kg/tds domperidone as treatment ,while the other group take the 0.4mg/kg/tds domperidone,0.6mg/kg/tds domperidone and the placebo respectively .

An objective index has been decided to evaluate the severity of feeding intolerance in the premature infant. 3kg/kg 5% glucose will be injected into the gastric tube .The residual glucose will be drawed out from the gastric tube. The residual percentage is the main result of the study.

The main result will be compared by the secondary result to help to explain the accuracy. The secondary result is the percentage of residual milk drawed out from the gastric tube from how many milk the infant take 3 hours ago.

Any adverse effect will be recorded and analysed to figure out whether is associate with the domperidone.

ELIGIBILITY:
Inclusion Criteria:

* the residual milk and glucose over 55%
* abdominal distention or vomiting;
* Reduce,delay or disruption of enteral feeding

Exclusion Criteria:

* Four weeks before the start of this study had participated in other clinical trials
* pulmonary hypertension;
* Infants with necrotizing enterocolitis
* Gastrointestinal tract malformation, congenital heart disease
* Pre-existing QT extend/between long QT syndrome;
* ascites
* Have been used or will use drugs suppress CYP3A4
* Other risk factors for prolong the QT

Ages: 20 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2015-11; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
the residual glucose percentage | 7 days
  3kg/kg 5% glucose will be injected into the gastric tube .The residual glucose will be drawed out from the gastric tube after 30 min

SECONDARY OUTCOMES:
the percentage of residual milk | 7 days
  the percentage of residual milk drawed out from the gastric tube from how many milk the infant take 3 hours ago.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: WeiMing Huang, professor, Study Chair — Nanfang Hosiptal
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No